CLINICAL TRIAL: NCT01314001
Title: Pharmacogenetics of Nicotine Addiction Treatment (PNAT)
Brief Title: Pharmacogenetics of Nicotine Addiction Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 811722; U01DA020830 (NIH)
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Nicotine Addiction
Keywords: Tobacco, Smoking, Varenicline, Nicotine Patch
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Varenicline; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Slow Metabolizers) (Placebo Comparator): Subjects in this arm are those identified as slow metabolizers of nicotine (based on their NMR) and will take placebo pills daily for twelve weeks & wear a placebo patch daily for eleven weeks.
  The placebo pill will look identical to the active varenicline tablets; however, they will not contain any active medication. Subjects will follow the same drug regimen as those in the active varenicline arm.
  The placebo patch will look identical to the active transdermal nicotine patches; however, they do not contain actual nicotine. Subjects will follow the same regimen as those in the active transdermal nicotine arm.
  All subjects in this arm will receive smoking cessation counseling during their sessions.
  Interventions: Drug: Placebo
- Varenicline (Slow Metabolizers) (Active Comparator): Subjects in this arm are those identified as slow metabolizers of nicotine (based on their NMR) and will take active varenicline pills daily for twelve weeks & wear a placebo patch daily for eleven weeks.
  When taking the active varenicline, subjects will follow the same treatment regimen per the manufacturer.
  The placebo patch will look identical to the active transdermal nicotine patches; however, they do not contain actual nicotine. Subjects will follow the same regimen as those in the active transdermal nicotine arm.
  All subjects in this arm will receive smoking cessation counseling during their sessions.
  Interventions: Drug: Varenicline
- Transdermal Nicotine (Slow Metabolizers) (Active Comparator): Subjects in this arm are those identified as slow metabolizers of nicotine (based on their NMR) and will take placebo pills daily for twelve weeks & will wear an active transdermal nicotine patch daily for eleven weeks.
  The placebo pill will look identical to the active varenicline tablets; however, they will not contain any active medication. Subjects will follow the same drug regimen as those in the active varenicline arm.
  When wearing the active transdermal nicotine, subjects will follow the same treatment regimen per the manufacturer.
  All subjects in this arm will receive smoking cessation counseling during their sessions.
  Interventions: Drug: Transdermal Nicotine
- Placebo (Normal Metabolizers) (Placebo Comparator): Subjects in this arm are those identified as normal metabolizers of nicotine (based on their NMR) and will take placebo pills daily for twelve weeks & wear a placebo patch daily for eleven weeks.
  The placebo pill will look identical to the active varenicline tablets; however, they will not contain any active medication. Subjects will follow the same drug regimen as those in the active varenicline arm.
  The placebo patch will look identical to the active transdermal nicotine patches; however, they do not contain actual nicotine. Subjects will follow the same regimen as those in the active transdermal nicotine arm.
  All subjects in this arm will receive smoking cessation counseling during their sessions.
  Interventions: Drug: Placebo
- Varenicline (Normal Metabolizers) (Active Comparator): Subjects in this arm are those identified as normal metabolizers of nicotine (based on their NMR) and will take active varenicline pills daily for twelve weeks & wear a placebo patch daily for eleven weeks.
  When taking the active varenicline, subjects will follow the same treatment regimen per the manufacturer.
  The placebo patch will look identical to the active transdermal nicotine patches; however, they do not contain actual nicotine. Subjects will follow the same regimen as those in the active transdermal nicotine arm.
  All subjects in this arm will receive smoking cessation counseling during their sessions.
  Interventions: Drug: Varenicline
- Transdermal Nicotine (Normal Metabolizers) (Active Comparator): Subjects in this arm are those identified as normal metabolizers of nicotine (based on their NMR) and will take placebo pills daily for twelve weeks & will wear an active transdermal nicotine patch daily for eleven weeks.
  The placebo pill will look identical to the active varenicline tablets; however, they will not contain any active medication. Subjects will follow the same drug regimen as those in the active varenicline arm.
  When wearing the active transdermal nicotine, subjects will follow the same treatment regimen per the manufacturer.
  All subjects in this arm will receive smoking cessation counseling during their sessions.
  Interventions: Drug: Transdermal Nicotine

INTERVENTIONS:
Drug: Varenicline — Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Other Names: Chantix
  Arms: Varenicline (Normal Metabolizers); Varenicline (Slow Metabolizers)
Drug: Placebo — Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Week 1 - 6: 21mg placebo patch Week 7 - 8: 14mg placebo patch Week 9 - 11: 7mg placebo patch
  Other Names: Placebo pills; Placebo patches
  Arms: Placebo (Normal Metabolizers); Placebo (Slow Metabolizers)
Drug: Transdermal Nicotine — Week 1-6: 21mg nicotine patch Week 7-8: 14mg nicotine patch Week 9-11: 7mg nicotine patch
  Other Names: Nicoderm CQ; Nicotine Patch
  Arms: Transdermal Nicotine (Normal Metabolizers); Transdermal Nicotine (Slow Metabolizers)

SUMMARY:
The purpose of this research program is to understand how a biomarker called the "nicotine metabolite ratio" (also referred to as NMR) may influence a smoker's ability to quit smoking.

DETAILED DESCRIPTION:
Smoking is an enormous public health problem with a great need for research to improve treatment outcomes. Our prior data indicates that the cytochrome P450 2A6 (CYP2A6) enzyme is critical in the metabolic inactivation of nicotine, and also influences smoking behavior and response to therapies. With a vision toward translation of our research to practice, we have characterized a genetically-informed biomarker of CYP2A6 activity, specifically the nicotine metabolite ratio (NMR; 3'hydroxycotinine/cotinine), which reflects both CYP2A6 genetic variation and environmental influences on CYP2A6 activity. The NMR is measured non-invasively in smokers with established reliability, stability, analytic validity, and efficacy as a predictor of the ability to quit smoking and treatment response in multiple retrospective trials. Translation of these findings to clinical practice requires validation in a prospective clinical trial comparing alternative therapies for smoking cessation. Thus, the proposed trial is a prospective, stratified, placebo-controlled, multi-center clinical trial of alternative therapies for smoking cessation treatment in approximately 1,200 smokers. Randomization to placebo (PLA), transdermal nicotine (TN), or varenicline (VAR) will be stratified prospectively based on the nicotine metabolite ratio (NMR). Abstinence from smoking at the end of treatment will be the primary outcome. Quit rate at 6-month follow-up is a secondary outcome. To facilitate translation to practice, analysis of the cost-effectiveness of our proposed approach will also be completed. The proposed research provides the next critical step to validate a genetically-informed diagnostic tool, the NMR, which clinicians can use in the future to optimize treatment decisions for their patients who wish to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be males and females

1. Between the ages of 18-65.
2. Smoke at least 10 cigarettes/day for the past 6 months.
3. Provide a baseline Carbon Monoxide (CO) reading greater than 10ppm at the Intake Session.
4. Are seeking smoking cessation treatment.
5. Plan to live in the area for the next 12 months.
6. Fluent English speaker.
7. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and Health Insurance Portability and Accountability Act (HIPAA) form. All subjects must consent to use a medically accepted method of birth control (e.g., condoms and spermicide, oral contraceptive, Depo-Provera injection, contraceptive patch, tubal ligation) or abstain from sexual intercourse during the time they are taking study medication (pills and patches) and for at least one month after the medication period ends. All female subjects of child-bearing potential should not be pregnant for the duration of the study.

Exclusion Criteria:

Smoking Behavior

1. Regular (daily) use of chewing tobacco, snuff or snus.
2. Current enrollment or plans to enroll in another smoking cessation or research program in the next 12 months.
3. Plan to use other nicotine substitutes or smoking cessation treatments in the next 12 months.
4. Provide a baseline CO reading less than or equal to 10ppm at the Intake Session.

Alcohol/Drug Exclusion Criteria

1. History (within the last year) or currently receiving treatment for substance abuse (e.g., alcohol, opioids, cocaine, marijuana, or stimulants), excluding nicotine.
2. Current use of cocaine and/or methamphetamines (urine drug screen at the Intake Session).
3. Current alcohol consumption that exceeds greater than 25 standard drinks/week.
4. Current alcohol abuse or dependence.
5. Current non-alcoholic psychoactive substance abuse or dependence.

Medical Exclusion Criteria

1. Women who are pregnant, planning a pregnancy, or lactating.
2. History of epilepsy or a seizure disorder.
3. Current medical problems for which transdermal nicotine is contraindicated including:

   * Allergy to latex.
   * History of kidney and/or liver disease, including transplant (self-report).
   * Uncontrolled hypertension (determined as a Systolic Blood pressure (SBP) reading greater than 160 and/or a Diastolic Blood Pressure (DBP) greater than 100).
4. Serious or unstable disease within the past 6 months.
5. History (last 6 months) of abnormal heart rhythms, tachycardia and cardiovascular disease (stroke, angina, heart attack) may result in ineligibility. These conditions will be evaluated on a case by case basis by the Study Physician.
6. Inability to provide a blood sample to be used to assess nicotine metabolite ratio.

Psychiatric Exclusion Criteria (as determined by self report & MINI)

1. Current diagnosis of major depression. Persons with a history of major depression, if stable for 6 months or longer, are eligible, provided they are not excluded based on medications (below).
2. Any suicide risk score on MINI or self-reported suicide attempt on telephone screen.
3. Current or past hypomanic/manic episode.
4. History or current diagnosis of Post Traumatic Stress Disorder (PTSD).
5. History or current diagnosis of psychotic disorder, bipolar disorder, schizophrenia.

Medication Exclusion Criteria

1. Current use or recent discontinuation (within the last 14-days) of:

   * Smoking cessation medication (e.g. Zyban, Wellbutrin, Wellbutrin SR, Chantix); NOTE: Once participants are found eligible for the study, they are instructed to use the smoking cessation medication provided to them by the study staff. If a subject reports an isolated (non-daily) instance of using a non-study smoking cessation medication, the study physician and PI will evaluate the situation and determine if it is safe for the subject to continue participation.
   * Anti-psychotic medications.
   * Certain medications used to treat depression, including Wellbutrin, Monoamine Oxidase Inhibitors (MAOIs), and tricyclic antidepressants.
   * Prescription stimulants (e.g. Provigil, Ritalin, Adderall).
2. Current use of:

   * Nicotine replacement therapy (NRT); NOTE: Once participants are found eligible for the study, they are told they should only use the NRT provided to them by the study staff. If a subject reports an isolated (non-daily) instance of NRT use during the study, they may be permitted to continue.
   * Tagamet (cimetidine).
   * Heart medications such as digoxin, quinidine, nitroglycerin; use of these medications may result in ineligibility and will therefore be evaluated on a case-by-case basis by the Study Physician.
   * Anti-coagulants (e.g., Coumadin, Warfarin).
3. Daily use of:

   * Opiate-containing medications for chronic pain; if a participant reports taking an opiate-containing medication every day for the 14 days prior to the telephone screen and/or Intake Session, the participant will be ineligible.
   * Rescue Inhalers (e.g. albuterol, proventil, ventolin, or maxair)

General Exclusion

1. Any medical condition, illness, disorder or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.
2. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, PhD, Principal Investigator — University of Pennsylvania; Rachel F Tyndale, PhD, Principal Investigator — University of Toronto
Locations (4):
- United States (3):
  - University at Buffalo - State University of New York, Buffalo, New York
  - Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, University of Texas, Houston, Texas
- Centre for Addiction and Mental Health, University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Tonkin SS, Betts JM, Dowd AN, Mahoney MC, Cinciripini PM, Schnoll RA, George TP, Tyndale RF, Hawk LW Jr. Daily Cigarette Abstinence and Smoking Rate With Varenicline: Relationships With Treatment, Craving, and Affect During the First Week of the Quit Attempt. Nicotine Tob Res. 2025 Nov 23;27(12):2328-2332. doi: 10.1093/ntr/ntaf095. PMID 40358028
- [Derived] Chenoweth MJ, Kim YJ, Nollen NL, Hawk LW Jr, Mahoney MC, Lerman C, Knight J, Tyndale RF. Genetic Prediction of Smoking Cessation Medication Side Effects: A Genome-Wide Investigation of Abnormal Dreams on Varenicline. Clin Pharmacol Ther. 2024 Jun;115(6):1277-1281. doi: 10.1002/cpt.3210. Epub 2024 Feb 19. PMID 38369951
- [Derived] Chenoweth MJ, Lerman C, Knight J, Tyndale RF. Influence of CYP2A6 Genetic Variation, Nicotine Dependence Severity, and Treatment on Smoking Cessation Success. Nicotine Tob Res. 2023 May 22;25(6):1207-1211. doi: 10.1093/ntr/ntac268. PMID 36789481
- [Derived] Tonkin SS, Colder C, Mahoney MC, Swan GE, Cinciripini P, Schnoll R, George TP, Tyndale RF, Hawk LW. Evaluating Treatment Mechanisms of Varenicline: Mediation by Affect and Craving. Nicotine Tob Res. 2022 Oct 26;24(11):1803-1810. doi: 10.1093/ntr/ntac138. PMID 35639828
- [Derived] Chenoweth MJ, Lerman C, Knight J, Tyndale RF. A Genome-Wide Association Study of Nausea Incidence in Varenicline-Treated Cigarette Smokers. Nicotine Tob Res. 2021 Aug 29;23(10):1805-1809. doi: 10.1093/ntr/ntab044. PMID 33713409
- [Derived] El-Boraie A, Chenoweth MJ, Pouget JG, Benowitz NL, Fukunaga K, Mushiroda T, Kubo M, Nollen NL, Sanderson Cox L, Lerman C, Knight J, Tyndale RF. Transferability of Ancestry-Specific and Cross-Ancestry CYP2A6 Activity Genetic Risk Scores in African and European Populations. Clin Pharmacol Ther. 2021 Oct;110(4):975-985. doi: 10.1002/cpt.2135. Epub 2021 Jan 1. PMID 33300144
- [Derived] Peng AR, Swardfager W, Benowitz NL, Ahluwalia JS, Lerman C, Nollen NL, Tyndale RF. Impact of early nausea on varenicline adherence and smoking cessation. Addiction. 2020 Jan;115(1):134-144. doi: 10.1111/add.14810. Epub 2019 Nov 5. PMID 31502736
- [Derived] Ashare RL, Thompson M, Leone F, Metzger D, Gross R, Mounzer K, Tyndale RF, Lerman C, Mahoney MC, Cinciripini P, George TP, Collman RG, Schnoll R. Differences in the rate of nicotine metabolism among smokers with and without HIV. AIDS. 2019 May 1;33(6):1083-1088. doi: 10.1097/QAD.0000000000002127. PMID 30946162
- [Derived] Robinson JD, Li L, Chen M, Lerman C, Tyndale RF, Schnoll RA, Hawk LW, George TP, Benowitz NL, Cinciripini PM. Evaluating the temporal relationships between withdrawal symptoms and smoking relapse. Psychol Addict Behav. 2019 Mar;33(2):105-116. doi: 10.1037/adb0000434. Epub 2019 Jan 7. PMID 30614717
- [Derived] Peng AR, Schnoll R, Hawk LW Jr, Cinciripini P, George TP, Lerman C, Tyndale RF. Predicting smoking abstinence with biological and self-report measures of adherence to varenicline: Impact on pharmacogenetic trial outcomes. Drug Alcohol Depend. 2018 Sep 1;190:72-81. doi: 10.1016/j.drugalcdep.2018.04.035. Epub 2018 Jun 26. PMID 29986268
- [Derived] Hamilton DA, Mahoney MC, Novalen M, Chenoweth MJ, Heitjan DF, Lerman C, Tyndale RF, Hawk LW Jr. Test-Retest Reliability and Stability of the Nicotine Metabolite Ratio Among Treatment-Seeking Smokers. Nicotine Tob Res. 2015 Dec;17(12):1505-9. doi: 10.1093/ntr/ntv031. Epub 2015 Mar 1. PMID 25732567
- [Derived] Lerman C, Schnoll RA, Hawk LW Jr, Cinciripini P, George TP, Wileyto EP, Swan GE, Benowitz NL, Heitjan DF, Tyndale RF; PGRN-PNAT Research Group. Use of the nicotine metabolite ratio as a genetically informed biomarker of response to nicotine patch or varenicline for smoking cessation: a randomised, double-blind placebo-controlled trial. Lancet Respir Med. 2015 Feb;3(2):131-138. doi: 10.1016/S2213-2600(14)70294-2. Epub 2015 Jan 12. PMID 25588294
- [Derived] Chenoweth MJ, Novalen M, Hawk LW Jr, Schnoll RA, George TP, Cinciripini PM, Lerman C, Tyndale RF. Known and novel sources of variability in the nicotine metabolite ratio in a large sample of treatment-seeking smokers. Cancer Epidemiol Biomarkers Prev. 2014 Sep;23(9):1773-82. doi: 10.1158/1055-9965.EPI-14-0427. Epub 2014 Jul 10. PMID 25012994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at four academic medical centers. From 11/16/2010 to 9/16/2013, participants were recruited through advertisements for a free smoking cessation program.
Pre-assignment Details: Subjects were randomly assigned to one of three treatment groups in a 1:1:1 ratio: "Placebo"; "Nicotine Patch"; or "Varenicline". Randomization was stratified by nicotine metabolite ratio - slow metabolizers of nicotine vs. normal metabolizers - and study site and blocked in blocks of 12 to maintain balance. Slow metabolizers were over-sampled.
Groups:
- Placebo (Slow Metabolizers): Slow metabolizers
  * Taking placebo pills daily for 12 weeks
  * Wearing placebo patches daily for 11 weeks
  * Received smoking cessation counseling during their sessions
- Placebo (Normal Metabolizers): Normal metabolizers
  * Taking placebo pills daily for 12 weeks
  * Wearing placebo patches daily for 11 weeks
  * Received smoking cessation counseling during their sessions
- Nicotine Patch (Slow Metabolizers): Slow metabolizers
  * Taking placebo pills daily for 12 weeks
  * Wearing active nicotine patches for 11 weeks (6 weeks of 21mg, 2 weeks of 14mg, 3 weeks of 7mg)
  * Received smoking cessation counseling during their sessions
- Nicotine Patch (Normal Metabolizers): Normal metabolizers
  * Taking placebo pills daily for 12 weeks
  * Wearing active nicotine patches for 11 weeks (6 weeks of 21mg, 2 weeks of 14mg, 3 weeks of 7mg)
  * Received smoking cessation counseling during their sessions
- Varenicline (Slow Metabolizers): Slow metabolizers
  * Taking active varenicline pills daily for 12 weeks (3 days of 0.5mg daily, 4 days of 0.5mg twice daily, and 77 days of 1mg twice daily)
  * Wearing placebo patches for 11 weeks
  * Received smoking cessation counseling during their sessions
- Varenicline (Normal Metabolizers): Normal metabolizers
  * Taking active varenicline pills daily for 12 weeks (3 days of 0.5mg daily, 4 days of 0.5mg twice daily, and 77 days of 1mg twice daily)
  * Wearing placebo patches for 11 weeks
  * Received smoking cessation counseling during their sessions
Period: Overall Study
Arm/Group | Placebo (Slow Metabolizers) | Placebo (Normal Metabolizers) | Nicotine Patch (Slow Metabolizers) | Nicotine Patch (Normal Metabolizers) | Varenicline (Slow Metabolizers) | Varenicline (Normal Metabolizers)
Started | 215 | 193 | 227 | 191 | 220 | 200
End-of-Treatment Visit | 156 | 141 | 179 | 146 | 174 | 160
6-Month Follow Up Survey | 146 | 137 | 165 | 135 | 157 | 139
Completed | 140 | 124 | 158 | 122 | 148 | 129
Not Completed | 75 | 69 | 69 | 69 | 72 | 71

BASELINE CHARACTERISTICS:
Population: The number of subjects who began treatment period in the project (intention-to-treat).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Slow Metabolizers) | Placebo (Normal Metabolizers) | Nicotine Patch (Slow Metabolizers) | Nicotine Patch (Normal Metabolizers) | Varenicline (Slow Metabolizers) | Varenicline (Normal Metabolizers) | Total
Number analyzed (Participants) | 215 | 193 | 227 | 191 | 220 | 200 | 1246
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11) | 47 (11) | 46 (11) | 46 (11) | 44 (12) | 46 (12) | 45 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 91 | 88 | 94 | 88 | 99 | 543
  Male | 132 | 102 | 139 | 97 | 132 | 101 | 703
Race/Ethnicity, Customized [Number; unit: participants]
  White | 97 | 128 | 117 | 119 | 99 | 133 | 693
  Black | 95 | 56 | 94 | 57 | 107 | 53 | 462
  Other | 23 | 9 | 16 | 15 | 14 | 14 | 91
Region of Enrollment [Number; unit: participants]
  Canada | 47 | 43 | 52 | 42 | 48 | 44 | 276
  United States | 168 | 150 | 175 | 149 | 172 | 156 | 970
Education level [Number; unit: participants] — Question on Demographics measure (self-report) completed at the Intake session ("What is the highest level of education you completed?").
  participants
    High school education or lower | 68 | 57 | 78 | 49 | 74 | 61 | 387
    Post-high school education | 147 | 136 | 149 | 142 | 146 | 139 | 859
Annual Income (US dollars) [Number; unit: participants] — Question on Demographics measure (self-report) completed at the Intake session ("What was your household income before taxes last year?").
  participants
    Greater than or equal to US$50,000 | 65 | 79 | 82 | 75 | 74 | 71 | 446
    Less than US$50,000 | 150 | 114 | 145 | 116 | 146 | 129 | 800
Employment Status [Number; unit: participants] — Question on Demographics measure (self-report) completed at the Intake session ("Are you currently employed full-time or part-time for salary or wages?").
  participants
    Not employed | 79 | 84 | 69 | 71 | 88 | 75 | 466
    Employed | 136 | 109 | 158 | 120 | 132 | 125 | 780
FTND Score [Mean (Standard Deviation); unit: units on a scale] — The Fagerstrom Test for Nicotine Dependence (FTND) is a six-item self-report scale that measures the level of nicotine dependence. Summary scores are calculated, ranging from 0 to 10, with higher scores indicating a greater difficulty quitting smoking.
  units on a scale | 5.3 (1.92) | 5.4 (2.00) | 5.2 (2.00) | 5.3 (1.89) | 5.1 (2.00) | 2.1 (2.02) | 5.2 (1.97)
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] — Self-report measure of the number of cigarettes smoked in a typical day.
  cigarettes per day | 17.6 (7.0) | 19.6 (8.7) | 17.6 (7.0) | 18.5 (7.0) | 16.7 (5.4) | 18.4 (6.3) | 18.0 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Quit Rate at End-of-Treatment (EOT)
Description: The percentage of ITT subjects who were verified as abstinent. Abstinence was defined as no self-reported smoking (not even a puff) for at least 7 days before the telephone assessment, with in-person verification for those self-reporting abstinence. In-person verification consisted of breath carbon monoxide analysis, with a reading of 8 parts-per-million or less confirming abstinence. Subjects who were lost to follow-up were considered smokers.
Time Frame: Week 11
Population: Intent-to-treat population (all subjects who received at least one dose of intervention).
Measure: Number; unit: percentage of ITT subjects
Arm/Group | Placebo (Slow Metabolizers) | Placebo (Normal Metabolizers) | Nicotine Patch (Slow Metabolizers) | Nicotine Patch (Normal Metabolizers) | Varenicline (Slow Metabolizers) | Varenicline (Normal Metabolizers)
Number analyzed (Participants) | 215 | 193 | 227 | 191 | 220 | 200
percentage of ITT subjects | 17.2 | 18.6 | 27.7 | 22.5 | 30.4 | 38.5

2. Secondary Outcome: 7-day Point Prevalence Quit Rate at 6-month Follow up Survey
Description: The percentage of ITT subjects who were verified as abstinent at the 6-month follow up survey. Abstinence was defined as no self-reported smoking (not even a puff) for at least 7 days before the telephone assessment, with in-person verification for those self-reporting abstinence. In-person verification consisted of breath carbon monoxide analysis, with a reading of 8 parts-per-million or less confirming abstinence. Subjects who were lost to follow-up were considered smokers.
Time Frame: Week 24
Population: Intent-to-treat population (all subjects who received at least one dose of intervention).
Measure: Number; unit: percentage of ITT subjects
Arm/Group | Placebo (Slow Metabolizers) | Placebo (Normal Metabolizers) | Nicotine Patch (Slow Metabolizers) | Nicotine Patch (Normal Metabolizers) | Varenicline (Slow Metabolizers) | Varenicline (Normal Metabolizers)
Number analyzed (Participants) | 215 | 193 | 227 | 191 | 220 | 200
percentage of ITT subjects | 14.4 | 12.9 | 21.6 | 13.6 | 19.1 | 22.0

3. Secondary Outcome: Total Side-Effect Severity Index at Pre-Quit
Description: The mean side-effect severity score by treatment group (placebo vs. nicotine patch vs. varenicline) and by NMR group (slow metabolizers vs. normal metabolizers).
  Side-effect severity was calculated using a Side Effects Checklists (SEC). 29 common side-effects associated with transdermal nicotine or varenicline treatment were rated by participants on a 0 (none) to 3 (severe) scale. For each participant at this timepoint, these scores were summed to calculate a total score, with a range of 0 to 87; a higher score indicated a higher severity of side-effects.
Time Frame: Pre-Quit (Week -1/Baseline)
Population: Intent-to-treat population (all subjects who received at least one dose of intervention).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Slow Metabolizers) | Placebo (Normal Metabolizers) | Nicotine Patch (Slow Metabolizers) | Nicotine Patch (Normal Metabolizers) | Varenicline (Slow Metabolizers) | Varenicline (Normal Metabolizers)
Number analyzed (Participants) | 215 | 193 | 227 | 191 | 220 | 200
units on a scale | 3.95 (4.84) | 3.40 (4.34) | 3.26 (3.97) | 3.97 (4.74) | 3.05 (3.93) | 3.57 (4.19)

4. Secondary Outcome: Total Side-Effect Severity Index at Target Quit Date
Description: as for outcome 3
Time Frame: Target Quit Date (Week 0)
Population: Intent-to-treat population (all subjects who received at least one dose of intervention).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Slow Metabolizers) | Placebo (Normal Metabolizers) | Nicotine Patch (Slow Metabolizers) | Nicotine Patch (Normal Metabolizers) | Varenicline (Slow Metabolizers) | Varenicline (Normal Metabolizers)
Number analyzed (Participants) | 215 | 193 | 227 | 191 | 220 | 200
units on a scale | 4.22 (4.37) | 4.27 (4.57) | 3.98 (3.59) | 4.28 (4.96) | 4.68 (4.66) | 4.06 (4.01)

5. Secondary Outcome: Total Side-Effect Severity Index at Week 1
Description: as for outcome 3
Time Frame: Week 1
Population: Intent-to-treat population (all subjects who received at least one dose of intervention).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Slow Metabolizers) | Placebo (Normal Metabolizers) | Nicotine Patch (Slow Metabolizers) | Nicotine Patch (Normal Metabolizers) | Varenicline (Slow Metabolizers) | Varenicline (Normal Metabolizers)
Number analyzed (Participants) | 215 | 193 | 227 | 191 | 220 | 200
units on a scale | 5.58 (5.08) | 5.46 (5.00) | 5.44 (5.03) | 5.58 (5.48) | 6.04 (5.23) | 5.26 (4.98)

6. Secondary Outcome: Total Side-Effect Severity Index at Week 4
Description: as for outcome 3
Time Frame: Week 4
Population: Intent-to-treat population (all subjects who received at least one dose of intervention).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Slow Metabolizers) | Placebo (Normal Metabolizers) | Nicotine Patch (Slow Metabolizers) | Nicotine Patch (Normal Metabolizers) | Varenicline (Slow Metabolizers) | Varenicline (Normal Metabolizers)
Number analyzed (Participants) | 215 | 193 | 227 | 191 | 220 | 200
units on a scale | 5.33 (5.70) | 4.93 (5.68) | 4.24 (4.40) | 4.52 (5.46) | 4.97 (4.88) | 4.39 (3.96)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the entire span of each subject's participation, which is approximately 1 year, 1 month (from initial phone screening to the 12-month follow up survey).
Description: Systematic Assessment: subjects completed a side effect checklist (SEC) during each study session over the course of the treatment period (target quit date through end-of-treatment). The SEC listed anticipated side effects that could be caused by the study medication. Subjects could also spontaneously report AEs at any time.
Arm/Group | Placebo (Slow Metabolizers) | Placebo (Normal Metabolizers) | Nicotine Patch (Slow Metabolizers) | Nicotine Patch (Normal Metabolizers) | Varenicline (Slow Metabolizers) | Varenicline (Normal Metabolizers)
Serious Adverse Events (participants affected / at risk) | 10/215 | 6/193 | 11/227 | 11/191 | 3/220 | 8/200
Other Adverse Events (participants affected / at risk) | 194/215 | 171/193 | 206/227 | 169/191 | 210/220 | 185/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Slow Metabolizers) (N=215) | Placebo (Normal Metabolizers) (N=193) | Nicotine Patch (Slow Metabolizers) (N=227) | Nicotine Patch (Normal Metabolizers) (N=191) | Varenicline (Slow Metabolizers) (N=220) | Varenicline (Normal Metabolizers) (N=200)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Episode of atrial fibrillation that required hospitalization
Heart Attack (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — Episodes of heart attack or heart attack-like symptoms
Diabetes diagnosis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Diagnosis made during hospitalization following heart attack-like symptoms
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Severe nausea/vomiting/abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Symptoms severe enough to require hospitalization.
Tongue Swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hospitalization due to swelling of the tongue
Death (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gall bladder issues (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hospitalized due to surgery or issues of the gall bladder
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Hospitalization due to pneumonia
Ankle injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Broken bones (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Broken bones due to accidents
Knee injuries (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — Knee injuries; may require surgery
Cancer; colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Diagnosis of colon cancer
Cancer; lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Diagnosis of lung cancer
Cancer; oral (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Diagnosis of oral cancer
Cancer; throat (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Diagnosis of throat cancer
Moderate cervical dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unknown whether benign or malignant
Seizures; cause unknown (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic Attacks (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep problems (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal thoughts (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Kidney stone procedure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COPD diagnosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hospitalization; COPD diagnosis
Severe asthma attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Required hospitalization
Abscess drainage; surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin/bone biopsy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Slow Metabolizers) (N=215) | Placebo (Normal Metabolizers) (N=193) | Nicotine Patch (Slow Metabolizers) (N=227) | Nicotine Patch (Normal Metabolizers) (N=191) | Varenicline (Slow Metabolizers) (N=220) | Varenicline (Normal Metabolizers) (N=200)
Chest Pain (Cardiac disorders) | 14 | 12 | 11 | 7 | 13 | 7
Heart Palpitations (Cardiac disorders) | 28 | 22 | 20 | 15 | 20 | 15
Irregular Heartbeat (Cardiac disorders) | 10 | 9 | 6 | 5 | 6 | 4
Abdominal Pain (Gastrointestinal disorders) | 22 | 19 | 31 | 22 | 43 | 29
Constipation (Gastrointestinal disorders) | 67 | 44 | 50 | 50 | 71 | 48
Diarrhea (Gastrointestinal disorders) | 32 | 45 | 30 | 24 | 38 | 24
Flatulence (Gastrointestinal disorders) | 82 | 77 | 85 | 69 | 94 | 81
Gas (Gastrointestinal disorders) | 110 | 101 | 108 | 91 | 111 | 98
Indigestion (Gastrointestinal disorders) | 50 | 42 | 45 | 36 | 50 | 54
Nausea (Gastrointestinal disorders) | 61 | 50 | 48 | 40 | 97 | 94
Vomiting (Gastrointestinal disorders) | 11 | 5 | 4 | 6 | 13 | 12
Dizziness (General disorders) | 28 | 28 | 26 | 16 | 39 | 19
Dry Mouth (General disorders) | 89 | 71 | 99 | 74 | 111 | 62
Fatigue (General disorders) | 73 | 71 | 88 | 65 | 88 | 79
Headache (General disorders) | 95 | 74 | 75 | 64 | 88 | 60
Body Weakness (Musculoskeletal and connective tissue disorders) | 9 | 9 | 7 | 8 | 20 | 6
Feel Weakness (Musculoskeletal and connective tissue disorders) | 36 | 37 | 41 | 32 | 45 | 30
Abnormal Dreams (Psychiatric disorders) | 68 | 64 | 94 | 88 | 97 | 89
Agitation (Psychiatric disorders) | 103 | 95 | 105 | 96 | 90 | 84
Anxiety (Psychiatric disorders) | 74 | 87 | 84 | 86 | 71 | 73
Depressed Mood (Psychiatric disorders) | 51 | 52 | 66 | 52 | 56 | 49
Disturbed Attention (Psychiatric disorders) | 54 | 50 | 46 | 47 | 53 | 40
Hostility (Psychiatric disorders) | 54 | 44 | 39 | 43 | 42 | 43
Insomnia (Psychiatric disorders) | 70 | 63 | 72 | 64 | 83 | 60
Irritability (Psychiatric disorders) | 125 | 123 | 130 | 119 | 128 | 114
Sleep Problems (Psychiatric disorders) | 109 | 81 | 103 | 100 | 118 | 109
Suicidal Thoughts (Psychiatric disorders) | 4 | 1 | 1 | 0 | 1 | 1
Skin Redness (Skin and subcutaneous tissue disorders) | 17 | 15 | 42 | 26 | 23 | 17
Skin Swelling/Rash (Skin and subcutaneous tissue disorders) | 23 | 21 | 25 | 23 | 30 | 14

LIMITATIONS AND CAVEATS:
A limitation is that few Hispanics or Asians were included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No